CLINICAL TRIAL: NCT02500576
Title: Phase II Study of MK-3475 in Conjunction With Lymphodepletion, TIL, and High or Low Dose IL-2 in Patients With Metastatic Melanoma
Brief Title: Pembrolizumab, Standard Chemotherapy, Tumor Infiltrating Lymphocytes, and High- or Low-Dose Aldesleukin in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0922; NCI-2015-01395 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0922 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Melanoma; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; Cyclophosphamide; fludarabine phosphate; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (pembrolizumab, high-dose aldesleukin) (Experimental): Patients receive standard lymphodepleting chemotherapy comprising cyclophosphamide IV over 2 hours on days -7 and -6 followed by fludarabine phosphate IVPB over 15-30 minutes on days -5 to -1. Patients also receive therapeutic tumor infiltrating lymphocytes IV over 15-60 minutes on day 0 followed by high-dose aldesleukin IV over 15 minutes every 8-16 hours for up to 15 doses on days 1-5. Beginning between 21-28 days after TIL infusion, patients receive maintenance therapy comprising pembrolizumab IV over 30 minutes every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Biological: Therapeutic Tumor Infiltrating Lymphocytes
- Arm II (pembrolizumab, low-dose aldesleukin) (Experimental): Patients receive standard lymphodepleting chemotherapy comprising cyclophosphamide and fludarabine phosphate and therapeutic tumor infiltrating lymphocytes as in Arm I, followed approximately 6 hours later by low-dose aldesleukin SC for 14 days. Patients also receive pembrolizumab as in Arm I.
  Interventions: Biological: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Quality-of-Life Assessment; Biological: Therapeutic Tumor Infiltrating Lymphocytes

INTERVENTIONS:
Biological: Aldesleukin — Given IV or SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine Phosphate — Given IVPB
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Therapeutic Tumor Infiltrating Lymphocytes — Given IV
  Other Names: Tumor Infiltrating Lymphocytes

SUMMARY:
This randomized phase II trial studies how well giving pembrolizumab with standard chemotherapy, tumor infiltrating lymphocytes (TIL), and aldesleukin works in treating patients with melanoma that has spread to other areas of the body. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide and fludarabine phosphate, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving an infusion of TIL, or white blood cells, may help stimulate the immune system to help kill more cells. Aldesleukin may also stimulate the white blood cells to kill melanoma cells. Giving pembrolizumab together with standard chemotherapy, TIL, and high- or low-dose aldesleukin may help stop the melanoma from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the overall response rates of pembrolizumab (MK-3475) combined with lymphodepletion, TIL and high or low dose aldesleukin (interleukin-2) therapy in patients with metastatic melanoma.

SECONDARY OBJECTIVES:

I. Comparison of progression free survival between the treatment arms. II. Comparison of overall survival between the treatment arms. III. Comparison of deep tumor responses (defined as over 60% reduction in tumor burden) between the treatment arms as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

IV. Number of complete responses in both treatment arms. V. Safety evaluations by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.

EXPLORATORY OBJECTIVES:

I. Identification of biomarkers predictive of treatment response or failure through immunohistochemistry, flow cytometry, gene expression changes as assessed by NanoString codeset, neo-antigen identification and complementary determining region (CDR)3 sequencing from blood and tumor samples acquired from baseline and on-treatment samples.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard lymphodepleting chemotherapy comprising of cyclophosphamide intravenously (IV) over 2 hours on days -7 and -6 followed by fludarabine phosphate IV piggyback (IVPB) over 15-30 minutes on days -5 to -1. Patients also receive therapeutic tumor infiltrating lymphocytes IV over 15-60 minutes on day 0 followed by high-dose aldesleukin IV over 15 minutes every 8-16 hours for up to 15 doses on days 1-5. Beginning between 21-28 days after TIL infusion, patients receive maintenance therapy comprising of pembrolizumab IV over 30 minutes every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive standard lymphodepleting chemotherapy comprising of cyclophosphamide, fludarabine phosphate, and therapeutic tumor infiltrating lymphocytes as in Arm I, followed approximately 6 hours later by low-dose aldesleukin subcutaneously (SC) once per day (QD) for 14 days. Patients also receive pembrolizumab as in Arm I.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* TURNSTILE I - SCREENING:
* Patients must have metastatic melanoma or stage III in-transit, subcutaneous, or regional nodal disease
* Patients must have a lesion amenable to resection for the generation of TIL on MD Anderson protocol 2004-0069
* Patients must receive a magnetic resonance imaging (MRI)/computed tomography (CT)/positron emission tomography (PET) of the brain within 6 months of signing informed consent; if new central nervous system (CNS) lesions are present, patient must have definitive treatment (including surgery or radiation); principal investigator (PI) or his designee should make final determination regarding enrollment
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 - 1 within 30 days of signing informed consent
* Patients previously treated with immunotherapy, targeted therapy, or no therapy (treatment naive) will be eligible
* Patients receiving cytotoxic agents will be evaluated by the PI or his designee for eligibility suitability
* Patients with a negative pregnancy test (urine or serum) must be documented within 14 days of screening for women of childbearing potential (WOCBP); a WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not had menses at any time in the preceding 12 consecutive months)
* TURNSTILE II - TREATMENT:
* Patients must sign the treatment consent document before Turnstile II screening procedures; before the treatment starts and at each visit, the patient will be asked to complete two quality of life questionnaires; It should take about 15 minutes to complete the questionnaires (Functional Assessment of Cancer Therapy General [FACT-G], FACT-Melanoma); patients must fulfill all of the following criteria to be eligible for Turnstile II of the study
* Patients must have adequate TIL that were previously harvested and then cryopreserved on MD Anderson Cancer Center (MDACC) protocol 2004-0069
* Patients who have had prior therapy (BRAF inhibitors, ipilimumab, anti PD-1 antibody or anti PD-L1 antibody) or treatment naive patients are eligible as long as toxicity from therapy is grade =< 1 or at baseline
* Patients must have at least one biopsiable measurable metastatic melanoma, lesion > 1 cm and must be amenable to undergoing serial biopsies through the course of therapy; this lesion must not be documented as one of the target lesions
* Patients may have central nervous system (CNS) metastases which have been treated and are radiographically stable for at least 4 weeks
* Patients of both genders must practice birth control for four months after receiving the preparative regimen (lymphodepletion) and continue to practice birth control throughout the study; patients must have a documented negative pregnancy test (urine or serum) for women who have menstruated in the past 12 months and without sterilization surgery
* Unless surgically sterile by bilateral tubal ligation or vasectomy of partner(s), or if the patient is post-menopausal, the patient agrees to continue to use a barrier method of contraception throughout the study such as: condom, diaphragm, hormonal, intrauterine device (IUD), or sponge plus spermicide; abstinence is an acceptable form of birth control
* Pregnancy testing will be performed within 14 days of screening for women of childbearing potential (WOCBP); a WOCBP has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 12 consecutive months (i.e. who has not had menses at any time in the preceding 12 consecutive months)
* Clinical performance status of ECOG 0-1 within 30 days of signing informed consent
* A stress cardiac test (stress thallium, stress multi-gated acquisition scan [MUGA], dobutamine echocardiogram or other stress test that will rule out cardiac ischemia) within 1 month of lymphodepletion
* 12-lead electrocardiogram (EKG) showing no active ischemia and corrected QT (QTc) interval less than 480 msec
* Pulmonary function tests (forced expiratory volume in 1 second [FEV1] > 65% or forced vital capacity [FVC] > 65% of predicted) within 1 month of lymphodepletion
* Have measurable disease based on RECIST 1.1 and immune related response (irRC) criteria
* Absolute neutrophil count (ANC) >= 1,500 /mcL (within 10 days of treatment initiation)
* Platelets >= 100,000 /mcL (within 10 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L (within 10 days of treatment initiation)
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 10 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN (within 10 days of treatment initiation) OR
* Direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN or =< 5 X ULN for subjects with liver metastases (within 10 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT)/activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* TURNSTILE I - SCREENING
* Active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system; PI or his designee shall make the final determination regarding appropriateness of enrollment
* Primary immunodeficiency and need for chronic steroid therapy, exception: patients on chronic physiological dose of steroid equivalent to prednisone < 10 mg/day is allowed
* Patients who are pregnant or nursing
* Presence of a significant psychiatric disease, which in the opinion of the principal investigator or his designee, would prevent adequate informed consent
* TURNSTILE II - TREATMENT
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiation of lymphodepletion; exception: patients on chronic physiologic dose of steroid equivalent to prednisone < 10 mg/day is allowed
* Has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to investigational or standard agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to lymphodepletion or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy, alopecia, hypophysitis stable on physiologic dose of steroid equivalent to prednisone < 10 mg/day, hypothyroidism stable on hormone replacement are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to initiation of lymphodepletion
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study; subjects with hypophysitis stable on physiologic dose of steroid will not be excluded from the study
* Has evidence of interstitial lung disease or has a history of non-infectious pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B virus HBsAg surface protein antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Any active systemic infections requiring intravenous antibiotics, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, such as abnormal stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease; PI or his designee shall make the final determination regarding appropriateness of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N Amaria, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A phase II randomized stuy for patients with lymphodepletion, ex-vivo expanded melanoma. Patients with prior surgical excission of a melanoma tumor from the outpatient clinic based on tumor size.
Pre-assignment Details: 18 participants consented and off-study; 16 participants treated, 1-participant was not eligible and not assigned an arm, 1-participant withdrew due to denial of insurance.
Groups:
- Arm 1-High Dose IL2: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion, Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0 TIL infusion; Day +1 - HD I2, 720,00IU/kg IV bolus q 8-16 hrs up to 15 doses, approx 12-16 hrs post T-cell Infusion; Day +22 MK-3475 200 mg IV
- Arm 2- Low Dose IL2: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion- Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0- TIL infustion; Da +1-+14: LD IL-2, 2 million IU SC bolus daily x 14 days approx 6 hrs post T-cell infusion; Day =22 MK-3475 200mg IV
Period: Overall Study
Arm/Group | Arm 1-High Dose IL2 | Arm 2- Low Dose IL2
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Death | 2 | 1
Not completed — Lack of Efficacy | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Those who were randomized
Groups:
- Arm 1- High Dose IL2: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion, Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0 TIL infusion; Day +1 - HD I2, 720,00IU/kg IV bolus q 8-16 hrs up to 15 doses, approx 12-16 hrs post T-cell Infusion; Day +22 MK-3475 200 mg IV
- Arm 2- High Dose IL2: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion- Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0- TIL infustion; Da +1-+14: LD IL-2, 2 million IU SC bolus daily x 14 days approx 6 hrs post T-cell infusion; Day =22 MK-3475 200mg IV
- Total: Total of all reporting groups
Arm/Group | Arm 1- High Dose IL2 | Arm 2- High Dose IL2 | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate in Each Arm
Description: The overall response rate will be computed separately by arm and presented with exact 95% confidence intervals. The overall response rate will be compared between the two treatment arms by using Fisher's exact test. The association between overall response rate and the same covariates will be assessed by using logistic regression.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion, Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0 TIL infusion; Day +1 - HD I2, 720,00IU/kg IV bolus q 8-16 hrs up to 15 doses, approx 12-16 hrs post T-cell Infusion; Day +22 MK-3475 200 mg IV
- Arm 2: 8 wks prior to screening- TIL harvest; 7 days prior to TIL infusion- Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0- TIL infustion; Da +1-+14: LD IL-2, 2 million IU SC bolus daily x 14 days approx 6 hrs post T-cell infusion; Day =22 MK-3475 200mg IV
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 7
Participants
  Partial Response | 1 | 1
  Stable Disease | 2 | 1
  Progressive Disease | 3 | 5
  Not Evaluable | 1 | 0

2. Secondary Outcome: Overall Survival
Description: The method of Kaplan and Meier will be used to estimate the distributions of overall survival and distributions will be compared between arms by using the log-rank test. Cox regression analysis will be used to assess the association between disease and clinical covariates of interest and overall survival.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 7
months | 9.7 [3 to NA] — The upper limit of the confidence interval is not estimable because of the small number of patients. | 8.8 [8.2 to NA] — The upper limit of the confidence interval is not estimable because of the small number of patients.

3. Secondary Outcome: Progression-free Survival
Description: The method of Kaplan and Meier will be used to estimate the distributions of progression-free survival, and distributions will be compared between arms by using the log-rank test. Cox regression analysis will be used to assess the association between disease and clinical covariates of interest and progression-free survival.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 7 | 7
months | 28.6 [8.9 to 92.2] | 14.3 [2.3 to 87.7]

4. Secondary Outcome: Change in Blood and Tumor Biomarkers
Description: A generalized linear mixed model approach to account for intra-patient correlation will be used to measure blood and tumor biomarkers collected over time.
Time Frame: Baseline and weeks 3, 6, and 9
Measure: Mean (Full Range); unit: ratio
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 4 | 7
ratio
  CD4/CD8 at Baseline | 1.96 [1.38 to 2.59] | 2.63 [1.03 to 4.01]
  CD4/CD8 at Day 21/Week 3 | 0.58 [0.21 to 1.11] | 0.52 [0.19 to 0.76]
  CD4/CD8 at Day 42/Week 6 | 0.75 [0.22 to 1.42] | 0.20 [0.10 to 0.27]
  CD4/CD8 at Week 9 | 0.58 [0.18 to 1.29] | 0.33 [0.15 to 0.79]
  CD8+/ T-reg at Baseline | 73.4 [18.0 to 205.8] | 37.19 [5.3 to 97.4]
  CD8+/ T-reg at Day 21/Week 3 | 10.2 [2.5 to 25.4] | 9.7 [1.8 to 43.4]
  CD8+/ T-reg at Day 42/Week 6 | 26.4 [2.5 to 67.1] | 30.2 [8.9 to 54.2]
  CD8+/ T-reg at Week 9 | 23.9 [2.8 to 36.6] | 91.6 [8.8 to 492.7]

ADVERSE EVENTS:
Time Frame: 7 years; 1 month
Groups:
- Arm 1- High Dose IL2: Lymphodepleting chemotherapy with fludarabine and cyclophosphamide; Day 0 TIL infusion; Day +1 - HD I2, 720,00IU/kg IV bolus q 8-16 hrs up to 15 doses, approx 12-16 hrs post T-cell Infusion; Day +22 MK-3475 200 mg IV
Arm/Group | Arm 1- High Dose IL2 | Arm 2- Low Dose IL2
All-Cause Mortality (participants affected / at risk) | 2/8 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1- High Dose IL2 (N=8) | Arm 2- Low Dose IL2 (N=8)
Death (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1- High Dose IL2 (N=8) | Arm 2- Low Dose IL2 (N=8)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 1 (1)
Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Activated Partioal thrombopllastin time prolonged (Investigations) | 6 (9) | 2
Adult Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alamine Aminotransferase Increased (Investigations) | 4 (10) | 3 (9)
Alkaline Phosphatase Increased (Investigations) | 4 (6) | 5 (16)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (13) | 5 (11)
Anemia (Blood and lymphatic system disorders) | 7 (60) | 6 (40)
Anorexia (Metabolism and nutrition disorders) | 7 (12) | 5 (9)
Anxiety (Psychiatric disorders) | 5 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 4 (8) | 5 (9)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (9)
Back Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bladder Spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Blood Bilirubin Increase (Investigations) | 3 (11) | 3 (8)
Blood Lymphatic System Disorder (Investigations) | 1 (2) | 0 (0)
Blurred Vision (Eye disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BHP (Renal and urinary disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 | 0 (0)
Cellulitis (Infections and infestations) | 1 | 1
Chest-Pain (Cardiac disorders) | 1 (1) | 0 (0)
Chills (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 4 (8)
CMV (Infections and infestations) | 0 (0) | 1 (1)
Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (9) | 5 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 4 (9)
CPK (Investigations) | 2 (2) | 0 (0)
Creatinine Increased (Investigations) | 3 (5) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dematitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetes Type 2 (Endocrine disorders) | 0 (0) | 2 (2)
Diaphoresis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 2 (6)
Diminished Breath Sounds (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Diminished Lung Sounds and Crackles (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Ecchymoses (Investigations) | 6 (9) | 4 (9)
Edema (generalized) (General disorders) | 1 (1) | 0
Edema Limbs (General disorders) | 3 (4) | 2 (2)
Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Eye Infection (Infections and infestations) | 0 | 1 (1)
Eye Pain (Eye disorders) | 0 | 4 (4)
Eye Redness (Eye disorders) | 0 | 1 (1)
Fatigue (General disorders) | 1 (1) | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (8) | 4 (8)
Fever (General disorders) | 3 (6) | 4 (9)
Flatulance (Social circumstances) | 1 | 0
Floaters (Investigations) | 1 (1) | 1 (1)
Fluid Retention (General disorders) | 1 (1) | 0
Flushing (Renal and urinary disorders) | 0 | 2 (3)
Fluid Overload (General disorders) | 1 (1) | 0
Gait Disturbance (General disorders) | 1 (1) | 0
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Generalized Edema (General disorders) | 2 (2) | 0 (0)
Gerneralized Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Generalized muscle weakness (General disorders) | 6 (9) | 6 (7)
Granulaoma Annulare (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Hayfever (General disorders) | 0 | 1 (2)
Head fullness (Nervous system disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 3 (5) | 3 (5)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Hematemsis (Gastrointestinal disorders) | 0 | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 1
Hemorrhodial Hemorrhage (General disorders) | 0 (0) | 1 (1)
Herpatic Pain (General disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Herpatic skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6) | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (5) | 4 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hyperthyrodism (Endocrine disorders) | 1 (1) | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (23) | 6 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (17) | 6 (16)
Hypokalemia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (4)
Hypomagnesenia (Metabolism and nutrition disorders) | 4 (5) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 5 (10) | 3 (5)
Hypotension (Vascular disorders) | 1 | 2 (2)
Hypothyrodism (Endocrine disorders) | 3 (3) | 2 (2)
Indigestion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1)
INR Increase (Investigations) | 6 (9) | 1 (1)
Insomnia (General disorders) | 5 (5) | 1 (2)
Iritis (Eye disorders) | 0 (0) | 1 (2)
Joint Range of Motion Decrease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (2)
Lip Infection (Infections and infestations) | 1 (1) | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0
Lynphedema (Vascular disorders) | 0 | 3 (3)
Lymphocyte Count Decrease (Investigations) | 2 (3) | 0
Malaise (General disorders) | 1 (1) | 0
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0
MRSA (Infections and infestations) | 1 (1) | 0
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle Weakness- lower limbs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Muscular Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Muscular Weakness- upper limbs (Musculoskeletal and connective tissue disorders) | 0 | 1 (3)
Myalgia (General disorders) | 3 (5) | 1 (1)
Myopathy (Cardiac disorders) | 1 (1) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Nausea (Gastrointestinal disorders) | 6 (12) | 5 (11)
Neutrophil Count decreased (Investigations) | 7 (26) | 7 (18)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7)
Non-Cardiac Chest Pain (Cardiac disorders) | 2 (2) | 2 (4)
Numbness (General disorders) | 0 | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Oral lesion (Gastrointestinal disorders) | 1 (1) | 0
Oral Thrush (Gastrointestinal disorders) | 0 | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Pain (generalized) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Pain (left side) (Musculoskeletal and connective tissue disorders) | 1 (4) | 0
Pain (left hip) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Pain (lower back) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Pain (right flank) (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (7) | 1 (1)
Pain ok skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pallor (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pericardial Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 2 (3)
Petechiae (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Phosphorus Level Increased (Metabolism and nutrition disorders) | 1 (1) | 0
Platelete Count Decreased (Investigations) | 7 (60) | 6 (36)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Pneumonia (Infections and infestations) | 1 (1) | 0
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (11) | 4 (6)
Race (face) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (6) | 2 (4)
Rash on Truck (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Seasonal Allergies (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Rhonchi (right and middle fields) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Right breast tenderness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Right toe pain (General disorders) | 0 | 1 (1)
Rigors (General disorders) | 1 (1) | 0
Seborrheic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sinus Bradycardia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus Pressure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Sinus Tachycardia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (6)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Sunburn (cheecks) (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0
Thrush (Gastrointestinal disorders) | 0 | 1 (1)
Tingling (bil feet) (Nervous system disorders) | 0 | 1 (1)
Tongue coated white (Gastrointestinal disorders) | 1 (1) | 0
Tremors (Bil hands) (Nervous system disorders) | 1 (1) | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0
Urinary Tract Infectins (Renal and urinary disorders) | 1 (1) | 1 (1)
Vaginal Yeast Infections (Reproductive system and breast disorders) | 1 (1) | 0
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0
Vitreous Hemorrhage (Eye disorders) | 1 (1) | 0
Volume Overload (General disorders) | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 3 (6) | 5 (10)
Watery Eyes (Eye disorders) | 1 (1) | 0
Weight Gain (Investigations) | 4 (5) | 1 (2)
Weight Loss (Investigations) | 3 (5) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0
White blood cell decreased (Blood and lymphatic system disorders) | 6 (20) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02500576/Prot_SAP_000.pdf